CLINICAL TRIAL: NCT01562431
Title: The Signal-Trial: Evaluation of a Screening Tool for Psychosocial Problems in Cancer Genetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: P11SIG; 2008-4016 (Other Grant/Funding Number: Dutch Cancer Society)
Record Dates: First submitted 2011-12-20; First posted 2012-03-23 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Psychosocial Issues; Cancer Genetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): Participants complete the Signal-checklist BUT counselors do not obtain the results of the checklist
  Interventions: Other: Feed-back
- Intervention (Other): Participants complete the Signal-checklist AND the counselor will get the results of the questionnaire
  Interventions: Other: Feed-back

INTERVENTIONS:
Other: Feed-back — Counselors will receive the results of the completed Signal-checklist completed by participants in the intervention group

SUMMARY:
Background

An important part of individuals undergoing genetic counseling and/or testing for cancer experience psychosocial problems and worries during or after this process. Approximately 20% of these individuals experience serious problems, such as fear for cancer in themselves or their relatives, family communication problems, unresolved grief, problems in coping with the DNA-test-results, difficulties in choices with regard to DNA-testing, preventive surgeries, and concerns about insurance or work. Research shows that these problems are frequently undetected by the counselors. Within the limited available time of a counseling session, a lot of information should be given to the counselee. This information is mostly biomedical and provider driven. Therefore psychosocial issues can be underexposed. The use of a brief questionnaire, completed by the counselee prior to the counseling session, can serve as a tool for the counselor to screen and address the relevant psychosocial issues in a systematic manner. Therefore, in 2009-2010 the investigators have developed and validated the 'Signal-checklist' to identify relevant psychosocial problems frequently encountered in the cancer-genetics setting, and need for extra psychosocial services. This 'Signal-checklist' can serve as a tool in screening systematically for psychosocial issues, addressing these issues and directing appropriate referrals to extra psychosocial services. The Signal-Trial will be performed to evaluate the use and effectiveness of the checklist.

Aim

The aim of the trial is to evaluate the implementation of a short, self-developed cancer-genetics checklist; the 'Signal-checklist', as an aid in 1) facilitating communication on psychosocial issues during the genetic counseling session, 2) increasing counselors awareness of psychosocial problems of the counselee, and 3) improving the management of these psychosocial problems during and after the process of genetic counselling.

Method

This study is a collaboration between the family cancer clinics of the NKI-AVL and the UMCU. Individuals requesting genetic counseling for the high incidence of cancer in their family are invited to participate in the trial. Participants will be asked to complete the 'Signal checklist' prior to their counseling visit. Participants (N=264) will be randomly assigned to one of the two study arms. The intervention group will receive feed-back on the 'Signal-checklist', whereas the control group will not receive feed-back. Three weeks after the DNA-test disclosure session, participants will be asked to complete again the 'Signal-checklist' followed by a telephone call by their counselor. Again, the results of the 'Signal-checklist' will be available to the counselor for participants in the intervention group, but not for the control group. Both the genetic counseling session and telephone call will be audio taped. Furthermore, all participants will be asked to complete three questionnaires on the Internet (or by mail, if preferred); 1) before randomization (3 weeks prior to the counseling session), 2) three weeks after the counseling session, and 3) four months after the potential DNA-test result disclosure. These questionnaires include items on communication during genetic counseling, the need for professional psychosocial support, cancer worries, satisfaction with received care, and experiences with the use of the 'Signal-checklist'. The audio-tapes and completed questionnaires will be used to measure psychosocial problems of the counselees, the awareness of the counselors of these problems, and the management of these problems. Secondary analysis will be conducted to assess the need for extra psychosocial services, satisfaction with genetic counseling, feasibility of implementing the 'Signal-checklist' and decreasing psychosocial problems over time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Sufficient command of the Dutch language to be able to complete questionnaires
* Attendees of a second visit at the family cancer clinic because of increased risk of developing cancer due to a hereditary predisposition

Exclusion Criteria:

* Those who do not fulfill the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Communication on psychosocial issues at the counseling session | 3 weeks after randomization
  The counseling session at the clinic will be audio taped, and content analyzed to evaluate counselor- counselee communication. A study-specific checklist will be used to rate whether psychosocial problems are discussed during the counseling session.
Counselors awareness of psychosocial problems of the counselee at the counseling session | 3 weeks after randomization
  After each consult with a counselee, the counselor will have to complete a short form regarding their awareness of psychosocial problems of the counselee. The level of agreement between the counselor and the counselee will be assessed
Management of these psychosocial problems of the counselee during the counseling session | 3 weeks after randomization
  Management of the psychosocial problems will be measured using the audio-taped sessions. The study-specific checklist will be used to rate whether problems are being counseled during the session and/or counselees are being referred to extra psychosocial services.
Communication on psychosocial issues at telephone follow-up | up to 4 months after randomization
  The telephone follow-up will be audio taped, and content analyzed to evaluate counselor- counselee communication. A study-specific checklist will be used to rate whether psychosocial problems are discussed during the counseling session.
Counselors awareness of psychosocial problems of the counselee at follow-up | Up to 4 months after randomization)
  After each consult with a counselee, the counselor will have to complete a short form regarding their awareness of psychosocial problems of the counselee. The level of agreement between the counselor and the counselee will be assessed
Management of these psychosocial problems of the counselee at follow-up | Up to 4 months after randomization
  Management of the psychosocial problems will be measured using the audio-taped sessions. The study-specific checklist will be used to rate whether problems are being counseled during the session and/or counselees are being referred to extra psychosocial services.

SECONDARY OUTCOMES:
Initiation of discussed problems | Counseling session (3 weeks after randomization) and telephone follow-up (up to 4 months after randomization)
Time spent on psychosocial problems | Counseling session (3 weeks after randomization) and telephone follow-up (up to 4 months after randomization)
Counselee and counselor's level of satisfaction | 4 weeks after counseling session (7 weeks after randomization) and 4 months after telephone follow-up (up to 8 months after randomization)
Levels of counselee cancer worries | Before randomization (Baseline, 1 week before randomization), 4 weeks after counseling session (7 weeks after randomization) and 4 months after telephone follow-up (up to 8 months after randomization)
Number of psychosocial problems | Counseling session (3 weeks after randomization) and telephone follow-up (up to 4 months after randomization) and 4 months after telephone follow-up (up to 8 months after randomization)
Counselee and counselor evaluation of the intervention/ feasibility of the implementation of the intervention | 4 weeks after counseling session (7 weeks after randomization) and 4 months after telephone follow-up (up to 8 months after randomization)

CONTACTS AND LOCATIONS:
Overall Officials: E.M.A. Bleiker, PHd., Principal Investigator — The Netherlands Cancer Institute; N.K. Aaronson, PHd., Principal Investigator — The Netherlands Cancer Institute; D.E.E. Hahn, MSc., Principal Investigator — The Netherlands Cancer Institute; I Kluijt, MSc., Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Eijzenga W, Aaronson NK, Kluijt I, Sidharta GN, Hahn DE, Ausems MG, Bleiker EM. The efficacy of a standardized questionnaire in facilitating personalized communication about problems encountered in cancer genetic counseling: design of a randomized controlled trial. BMC Cancer. 2014 Jan 15;14:26. doi: 10.1186/1471-2407-14-26. PMID 24428912